CLINICAL TRIAL: NCT05931172
Title: Comparative Effects of Dual Task and Proprioceptive Neuromuscular Facilitation on Balance ,Cognition and Motor Function in Chronic Stroke Patients
Brief Title: Comparative Effects of Dual Task and PNF on Balance ,Cognition and Motor Function in Chronic Stroke Patients .
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/LHR/23/0224 nadia
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Stroke
Keywords: chronic stroke; PNF; Dual task; Hemiplegia
MeSH Terms: conditions — Stroke; Hemiplegia | interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual tasking (Experimental): Dual tasking utilizes a task-specific approach to balance training, applying repeated exposure to unpredictable mechanical perturbations that mimic balance disturbances experienced in daily life.
  Interventions: Other: Dual tasking
- Proprioceptive neuromuscular facilitation (Experimental): Proprioceptive neuromuscular facilitation (PNF) is a therapeutic approach that uses cutaneous, proprioceptive and auditory input to produce functional improvement in motor output.
  Interventions: Other: PNF(proprioceptive neuromuscular facilitation exercises)

INTERVENTIONS:
Other: Dual tasking — Dual-task training is an emerging task-specific intervention that aims to improve reactive balance control after destabilizing perturbations in a safe and controlled environment. Dual tasking is given by therapist in unexpected directions to challenge patients reactive balance. In this study dual tasking will be given manually and on hurdles.
  Daily 45 mins of exercise sessions of dual-task training like walking with talking , walking with a filled cup of water, walking with looking on clock performed for total eight weeks and 5 days a week.
  Arms: Dual tasking
Other: PNF(proprioceptive neuromuscular facilitation exercises) — PNF involves both stretching and contracting (activation) of the muscle group being targeted in order to achieve maximum static flexibility, along with its D1&D2 flexion/extension patterns to improve dynamic flexibility and thus improving balance and coordination.
  total 8 weeks session will be given to patients. 45 mins session/each day for 5 days a week.
  Arms: Proprioceptive neuromuscular facilitation

SUMMARY:
The aim of this study is to compare the effect of dual tasking and proprioceptive neuromuscular facilitation on balance, cognition and motor function in chronic stroke patients. It will be randomized clinical trial.

DETAILED DESCRIPTION:
Stroke is the major cause of disability and mortality worldwide. A stroke is defined as an abrupt neurological outburst caused by impaired perfusion through the blood vessels to the brain. Every year the number of patients affected by stroke is rising thereby putting extra pressure on socioeconomic conditions in developing countries. Major complications of stroke include hemiplegia leading to upper limb dysfunction along with gait abnormalities. This study will be conducted to determine the effects of proprioceptive neuromuscular facilitation exercises versus dual-task training on balance, cognition, and motor function in chronic stroke patients. The randomized clinical trial will be conducted, participants will be selected through Non-probability convenience sampling technique and then randomly allocated into two treatment groups.

ELIGIBILITY:
Inclusion Criteria:

item

* Both male and female
* Age 50-70 years.
* Person should be able to walk 10meter distance with or without assistance.
* Patient should be Cognitively able to perform required task.
* Chronic Stroke patients with strength >2 on manual muscle testing.

Exclusion Criteria:

item

* Any Gait impairment .
* Patients with comorbidities like cardiac pathologies.
* Patients with dementia .
* History of fall in last 6 months.
* History of Severe Freezing episodes.
* History of Camptocormia (axial deformity.
* Central or peripheral paresis.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-02-25 (Actual); Primary Completion 2023-10-18 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Berg balance scale | 8th week
  Berg balance scale is used to find and access the balance issues. This scale consists of 14 task which related to everyday life. Each function rates from 0 (worst) to 4 (best) along a dependence and independence sequence. In this test, we gradually reduce the base of support from sitting and standing to single-leg stance, assess a subject's capacity to sustain positions or movements of increasing difficulty. One's ability to change position is also evaluated(
Montreal Cognitive Assessment (MoCA) Scale | 8th week
  MoCA scale is used to meaured cognition .Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform,
  1=performs partially and 2=performs fully. The total possible scale score is 226.
Fugal meyer assessment scale | 8th week
  The Fugl-Meyer Assessment of Lower Extremity (FMA-LE) is a widely used and recommended scale for evaluation of post-stroke motor impairment. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.
  The scale is comprised of five domains and there are 155 items in total

CONTACTS AND LOCATIONS:
Overall Officials: hira jabeen, Principal Investigator — Riphah International University
Locations (1):
- CIVIL Hospital, Chak Four Hundred Fifty-four, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kuriakose D, Xiao Z. Pathophysiology and Treatment of Stroke: Present Status and Future Perspectives. Int J Mol Sci. 2020 Oct 15;21(20):7609. doi: 10.3390/ijms21207609. PMID 33076218
- [Background] Nguyen PT, Chou LW, Hsieh YL. Proprioceptive Neuromuscular Facilitation-Based Physical Therapy on the Improvement of Balance and Gait in Patients with Chronic Stroke: A Systematic Review and Meta-Analysis. Life (Basel). 2022 Jun 13;12(6):882. doi: 10.3390/life12060882. PMID 35743913
- [Background] Belas Dos Santos M, Barros de Oliveira C, Dos Santos A, Garabello Pires C, Dylewski V, Arida RM. A Comparative Study of Conventional Physiotherapy versus Robot-Assisted Gait Training Associated to Physiotherapy in Individuals with Ataxia after Stroke. Behav Neurol. 2018 Feb 20;2018:2892065. doi: 10.1155/2018/2892065. eCollection 2018. PMID 29675114
- [Background] Hernandez ED, Forero SM, Galeano CP, Barbosa NE, Sunnerhagen KS, Alt Murphy M. Intra- and inter-rater reliability of Fugl-Meyer Assessment of Lower Extremity early after stroke. Braz J Phys Ther. 2021 Nov-Dec;25(6):709-718. doi: 10.1016/j.bjpt.2020.12.002. Epub 2020 Dec 17. PMID 33358073
- [Background] Villepinte C, Catella E, Martin M, Hidalgo S, Techene S, Lebely C, Castel-Lacanal E, de Boissezon X, Chih H, Gasq D. Validation of French upper limb Erasmus modified Nottingham Sensory Assessment in stroke. Ann Phys Rehabil Med. 2019 Jan;62(1):35-42. doi: 10.1016/j.rehab.2018.03.004. Epub 2018 Apr 13. PMID 29660413
- [Background] Bergmann J, Krewer C, Muller F, Jahn K. A new cutoff score for the Burke Lateropulsion Scale improves validity in the classification of pusher behavior in subactue stroke patients. Gait Posture. 2019 Feb;68:514-517. doi: 10.1016/j.gaitpost.2018.12.034. Epub 2018 Dec 26. PMID 30623845